CLINICAL TRIAL: NCT05752682
Title: Guideline-based Global Approach to the Management of Faints and Falls in a Dedicated Outpatient Facility
Brief Title: Global Approach to Faint and Falls
Acronym: F2
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Michele Brignole, Principal Investigator, Istituto Auxologico Italiano
Other Study IDs: 09C021
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Syncope; Fall
Keywords: Syncope; Fall; Tilt table test; Ambulatory blood pressure monitoring; carotid sinus massage; implantable loop recorder; Treatment; Diagnosis
MeSH Terms: conditions — Syncope; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Syncope and fall: Consecutive patients aged ≥40 years referred to the Faint & Fall Clinics for assessment of an episode of faint or fall.
  Interventions: Diagnostic Test: Diagnostic pathway

INTERVENTIONS:
Diagnostic Test: Diagnostic pathway — Each included patient will undergo to the faint and fall protocol, to assess the effectiveness of a patients' flow pathways developed in accordance with the most recent guidelines on syncope of the European Society of cardiology and of guidelines on falls of the American and British Geriatrics Societies.

SUMMARY:
Syncope is the most frequent cause of transient loss of consciousness. Falls are very common in older people. If the falls are unexplained and not accidental, it is likely that the patient had a syncope event and showed a lack of awareness for loss of consciousness. The management of unexplained falls is the same as that of syncope. There is a gap between the best available scientific evidence provided by the guidelines and the need to disseminate these concepts in clinical practice. The absence of a systematic comprehensive approach to fainting and falls results in higher health and social costs, unnecessary hospitalizations and diagnostic procedures, prolonged hospital stays, lower diagnostic rates, and higher rates of misdiagnosis and symptomatic recurrence.

Aim of the study The aim of the study is to assess the efficacy (adherence) of a diagnostic protocol and the costs of a comprehensive guideline-based approach to the management of fainting and falls in a population of consecutive patients referred to a dedicated multidisciplinary outpatient facility.

Primary endpoint:

1. Prevalence rate of patients with unexplained fall undergoing diagnostic investigations for syncope among those initially subjected to a diagnostic evaluation for falls.

Secondary endpoints:

1. Comparison between patients initially assigned to syncope and those assigned to unexplained fall in terms of diagnostic tests and final diagnosis.
2. Comparison between patients initially assigned to syncope and those assigned to unexplained fall in terms of adherence to guideline recommendations.
3. Analysis of costs per patient of fall and syncope protocols
4. All previous analyses will be performed according to the following age groups: ≥75, 74-65 and 64-40 years.

Inclusion criteria

1. Consecutive patients >40 years of age, belonging to the Cwithin Fainting and Falls for the evaluation of an episode of syncope or fall.
2. Fragile patients at risk of falling.

Exclusion criteria:

1. Patients aged <40 years
2. Patients with dental falls
3. Patients with a known diagnosis of syncope
4. Patients in whom syncope and fall are secondary symptoms of severe underlying comorbidities

DETAILED DESCRIPTION:
1. Background. Syncope is the most frequent cause of transient loss of consciousness. Falls are very common in older people. If the falls are unexplained and not accidental, it is likely that the patient had a syncope event and showed a lack of awareness for loss of consciousness. The management of unexplained falls is the same as that of syncope. There is a gap between the best available scientific evidence provided by the guidelines and the need to disseminate these concepts in clinical practice. The absence of a systematic comprehensive approach to fainting and falls results in higher health and social costs, unnecessary hospitalizations and diagnostic procedures, prolonged hospital stays, lower diagnostic rates, and higher rates of misdiagnosis and symptomatic recurrence.
2. Aims of the study.

   To assess the effectiveness (adherence) of a patient flow pathway and cost of a guideline-based global approach to the management of faints and falls in patients referred to dedicated multidisciplinary outpatient facilities. We will considerer the following endpoints:

   Primary-endpoint:

   I. Point and interval prevalence estimation of patients with unexplained falls among those who underwent fall diagnostic assessment at initial presentation and then moved to faint pathway for prosecution of diagnostic assessment and its determinants.

   Secondary endpoints:

   I. Point and interval estimate of the agree proportion between initial presentation and final diagnosis in patients initially assigned to faint and those with unexplained falls.

   II. Descriptive comparison between patients initially assigned to faint and those with unexplained falls in terms of diagnostic assessment and adherence rate to the recommendations of the guidelines

   III. Descriptive cost analysis of the faint and fall protocol (costs of investigations per patient).

   Moreover, all previous analysis will be performed also for predefined age subgroups (≥75, 74-65 and 64-40 years).
3. Study design Prospective observational study

Inclusion criteria

- Consecutive patients aged ≥40 years referred to the Faint & Fall Clinics for assessment of an episode of faint or fall. The patients will be recruited from the second half of 2020 and the recruitment will continue until to the achievement of the sample size

Exclusion criteria:

* Patients with age <40 years
* Patients with incidental fall
* Patients with an established diagnosis of syncope
* Patients in whom syncope and fall are secondary symptoms of severe underlying comorbidities (e.g: acute myocardial infarction, pulmonary embolism, acute haemorrage)

Patients' flow Each included patient will undergo to the faint and fall protocol, to assess the effectiveness of a patients' flow pathways (shown in the figure 1) developed in accordance with the most recent guidelines on syncope of the European Society of cardiology (1) and of guidelines on falls of the American and British Geriatrics Societies (2). The detailed flow pathway is described in the Appendix.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged ≥40 years referred to the Faint & Fall Clinics for assessment of an episode of faint or fall.

Exclusion Criteria:

* Patients with age <40 years
* Patients with incidental fall
* Patients with an established diagnosis of syncope
* Patients in whom syncope and fall are secondary symptoms of severe underlying comorbidities (e.g: acute myocardial infarction, pulmonary embolism, acute haemorrage)

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with faint or fall referred to a Syncope Unit for diagnosis and therapy
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Unexplained falls | 1 year
  Point and interval prevalence estimation of patients with unexplained falls, among those who underwent fall diagnostic assessment at initial presentation and then moved to faint pathway for prosecution of diagnostic assessment and its determinants.

SECONDARY OUTCOMES:
Final diagnosis | 1 year
  Point and interval estimate of the agree proportion between initial presentation and final diagnosis in patients initially assigned to faint and those with unexplained falls.
Comparison | 1 year
  Descriptive comparison between patients initially assigned to faint and those with unexplained falls in terms of diagnostic assessment and adherence rate to the recommendations of the guidelines
Costs | 1 year
  Descriptive cost analysis of the faint and fall protocol (costs of investigations per patient).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Background] Panel on Prevention of Falls in Older Persons, American Geriatrics Society and British Geriatrics Society. Summary of the Updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011 Jan;59(1):148-57. doi: 10.1111/j.1532-5415.2010.03234.x. PMID 21226685

DOCUMENTS (1):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT05752682/Prot_000.pdf